CLINICAL TRIAL: NCT03044730
Title: Phase II Study of Pembrolizumab and Capecitabine for Advanced Triple Negative and Hormone-Refractory Breast Cancer
Brief Title: Pembrolizumab and Capecitabine in Treating Patients With Locally Advanced or Metastatic Triple Negative or Hormone-Refractory Breast Cancer That Cannot Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Gradishar, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16B08; STU00203215 (CTRP (Clinical Trial Reporting Program)); NU 16B08 (Other: Northwestern University); P30CA060553 (NIH); NCI-2017-00152 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Estrogen Receptor Negative; HER2/Neu Negative; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Capecitabine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, capecitabine) (Experimental): Patients receive pembrolizumab IV on day 1 and capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
The purpose of this study is to see whether a combination of two different drugs - pembrolizumab and capecitabine - is safe, and if it might be effective in treating triple negative and hormone-refractory breast cancer. Pembrolizumab is a type of drug that contains an antibody. Antibodies are the part of your immune system that finds things that don't belong in your body, such as bacteria or viruses. The antibody in pembrolizumab finds and blocks a protein, which allows your immune system to target and destroy cancer cells. Pembrolizumab is Food and Drug Administration (FDA) approved for other types of cancer. It is not approved for breast cancer, meaning that it is an "experimental" or "investigational" treatment. Capecitabine is a type of chemotherapy pill that is a standard treatment and FDA-approved for breast cancer. It stops the cancer cells from being able to multiply.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the median progression-free survival (median PFS) for participants receiving pembrolizumab with capecitabine for the treatment of locally advanced or metastatic triple negative breast cancer (TNBC) and hormone-refractory metastatic breast cancer (MBC).

SECONDARY OBJECTIVES:

I. To describe the objective response rate (ORR) for participants receiving pembrolizumab with capecitabine for the treatment of locally advanced or metastatic TNBC and hormone-refractory MBC.

II. To describe the safety and tolerability of the combination of pembrolizumab and capecitabine for the treatment of locally advanced or metastatic TNBC and hormone-refractory MBC.

TERTIARY OBJECTIVES:

I. Analysis of expression of programmed cell death 1 ligand 1 (PD-L1) through immunohistochemical (IHC) analysis.

II. To assess circulating tumor DNA (ctDNA). III. To evaluate ORR and median-PFS using immune-related Response Evaluation Criteria in Solid Tumors (irRECIST).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) on day 1 and capecitabine orally (PO) twice daily (BID) on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed unresectable, locally advanced or metastatic breast cancer that meets one of the following:

  * Triple negative, defined as estrogen receptor (ER) negative, progesterone receptor (PR) negative, human epidermal growth factor receptor 2 (HER2) negative; HER2 negative defined as immunohistochemistry (IHC) 0 or 1+ or fluorescence in situ hybridization (FISH) negative
  * Hormone-refractory breast cancer which denotes progression to endocrine therapy (e.g., tamoxifen, aromatase inhibitors, fulvestrant) unless contraindicated
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have a life expectancy of >= 90 days
* Patients must have baseline laboratory tests within the following parameters at least 4 weeks (28 days) prior to registration:
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Females of child-bearing potential (FOCBP) must have a negative serum or urine pregnancy test within 7 days prior to registration and must be at least within 3 days prior to first dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * (Note: a FOCBP is any woman [regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice] who meets the following criteria:
  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Female subjects of childbearing potential (FOCBP) must be willing to use an adequate method of contraception; contraception must be used for the course of the study through 120 days after the last dose of study medication

  * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception; contraception must be used starting with the first dose of study therapy through 120 days after the last dose of study therapy

  * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study
* Patients must be willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Patient must be able to swallow and retain oral medication

Exclusion Criteria:

* Patients with documented HER2-positive metastatic disease are not eligible, even if their primary breast cancer was HER2-negative
* Patients who have received prior anti-cancer therapy (e.g., biologic or other targeted therapy, chemotherapy) within 2 weeks prior to registration; hormone therapy is permitted until registration

  * Note: patients who received prior anti-PD-1, PD-L1 or PD-L2 agents are still eligible
* Patients who have not recovered from adverse events to grade 1 severity or lower due to agents administered more than 2 weeks earlier than registration, are not eligible, except for stable sensory neuropathy (=< grade 2) and alopecia
* Patients who have received radiotherapy =< 4 weeks prior to registration, with the exception of palliative radiotherapy, who have not recovered from side effects of such therapy to baseline or grade =< 1 are not eligible for participation
* Patients with central nervous system (CNS) involvement may participate if they meet all the following criteria:

  * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment,
  * Clinically stable with respect to the CNS tumor at the time of screening
* Patients who have undergone major surgery =< 4 weeks prior to registration or have not recovered from side effects of such procedure are not eligible for participation
* Patients may not be receiving any other investigational agents
* Patients who have a history of allergic reactions or hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab and/or humanized antibodies are not eligible
* Known hypersensitivity to capecitabine, fluorouracil, or any component of the formulation

  * Note: prior capecitabine is permitted
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis or glomerulonephritis

  * Patients with history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study
  * Patients with controlled type I diabetes mellitus on a stable dose of insulin regimen for more than a month may be eligible for this study
* Patients who have evidence of active, noninfectious pneumonitis or have a history of severe pneumonitis that required treatment with steroids are not eligible for this study; (Note: replacement physiologic dose of steroids [prednisone 10 mg daily or equivalent] are allowed)
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension that is not controlled on medication (defined as >= 140/100 at rest, average of 3 consecutive readings)
  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Clinically significant electrocardiogram (ECG) abnormality, e.g., a repeated demonstration of a QTc interval > 500 ms
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Known positive test for human immunodeficiency virus (HIV)
  * Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
  * Active tuberculosis
  * Prior allogeneic bone marrow transplantation or solid organ transplant
  * Administration of a live, attenuated vaccine within 4 weeks before starting the study treatment or anticipation that a live attenuated vaccine will be required during the study
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing (lactating) are not eligible
* Patients exhibiting any other condition that would, in the Investigator's judgment, preclude patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures are not eligible for participation; this might include, but is not limited to, infection/inflammation, intestinal obstruction, and/or social/psychological complications
* Patients with impaired gastrointestinal (GI) function or GI disease that may significantly alter absorption of oral capecitabine (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) are not eligible for participation
* Patients with a history of another malignancy that progressed or required treatment within 5 years prior to registration are not eligible for participation; Note: the exceptions to this include non-melanoma skin cancer or excised carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2021-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sarika Jain, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Northwestern Lake Forest Hospital, Lake Forest, Illinois

REFERENCES:
- [Derived] Shah AN, Flaum L, Helenowski I, Santa-Maria CA, Jain S, Rademaker A, Nelson V, Tsarwhas D, Cristofanilli M, Gradishar W. Phase II study of pembrolizumab and capecitabine for triple negative and hormone receptor-positive, HER2-negative endocrine-refractory metastatic breast cancer. J Immunother Cancer. 2020 Feb;8(1):e000173. doi: 10.1136/jitc-2019-000173. PMID 32060053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for enrollment on May 25th, 2017 with an accrual goal of 30 patients. The first patient started treatment on May 30th, 2017. The study closed permanently to further enrollment on March 12th, 2018 as the accrual goal was met.
Groups:
- Treatment: Pembrolizumab + Capecitabine: This is a single-arm, phase II study of patients with triple negative (TN) or hormone receptor-positive endocrine-refractory (HR+) metastatic breast cancer (MBC) who were candidates for capecitabine. Patients were treated with pembrolizumab 200 mg intravenously day 1 and capecitabine 1000 mg/m2 by mouth twice daily on days 1-14 of a 21-day cycle. Patients continued treatment until disease progression or unacceptable toxicity. After discontinuation of study drugs, patients were assessed every 3 months up to 2 years for PFS, with visits and/or phone calls.
Period: 3 Cycles of Pembro + Capecitab
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Started | 30
Attempted Cycle 1 | 30
Attempted Cycle 2 | 28
Attempted Cycle 3 | 26
Completed | 26
Not Completed | 4
Not completed — Progressive Disease | 1
Not completed — Patient non-compliant with capecitabine | 1
Not completed — Death | 1
Not completed — Adverse Event | 1
Period: Cycles 4 and Beyond
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Started | 26
Assessed for Cycle 4 | 26
Started Cycle 4 | 20
Went on to Cycle 5 and Beyond | 16
Completed | 16
Not Completed | 10
Not completed — Progressive Disease | 9
Not completed — Adverse Event | 1
Period: On Follow-up for 2 Years
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Started (Pts who received at least 1 cycle of treatment go in follow-up. One pt is still on treatment.) | 29
Completed | 4
Not Completed | 25
Not completed — Still in follow-up | 7
Not completed — Lost to Follow-up | 1
Not completed — Death | 17

BASELINE CHARACTERISTICS:
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30
Triple Negative vs Hormone Receptor Positive MBC [Count of Participants; unit: Participants] — Patients on study must have histologically-confirmed unresectable, locally advanced or metastatic breast cancer (MBC) that meets one of the following:
  • Triple negative (TN), defined as estrogen receptor (ER) negative, progesterone receptor (PR) negative, human epidermal growth factor receptor 2 (HER2) negative.
  or
  • HER2- negative hormone-refractory breast cancer which denotes progression on one or more endocrine therapies (e.g., tamoxifen, aromatase inhibitors, fulvestrant) unless contraindicated (referred to as Hormone Receptor Positive, or HR+).
  Participants
    Triple Negative MBC | 16
    Hormone Receptor Positive MBC | 14

OUTCOME MEASURES:

1. Primary Outcome: Median PFS (Median Progression-Free Survival)
Description: To evaluate the median Progression-Free Survival (PFS) for participants receiving pembrolizumab with capecitabine for the treatment of locally advanced or metastatic TNBC and hormone-refractory MBC. PFS is defined as the length of time during and after the treatment that a patient does not experience progression.
  Progressive Disease (PD) as defined per RECIST 1.1 is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  PFS was analyzed using a Kaplan-Meier curve.
  For PFS, assumptions were that the addition of pembrolizumab would increase PFS to 5 months compared to historical control of 3 months.
Time Frame: Approximately 20 months
Population: One patient was not evaluable due to non-compliance with capecitabine. Three patients were not evaluable because they did not reach 3 cycles of treatment (per Protocol).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment: Pembrolizumab + Capecitabine: This is a single-arm, phase II study of patients with triple negative (TN) or hormone receptor-positive endocrine-refractory (HR+) metastatic breast cancer (MBC) who were candidates for capecitabine. Patients were treated with pembrolizumab 200 mg intravenously day 1 and capecitabine 1000 mg/m2 by mouth twice daily on days 1-14 of a 21-day cycle. Patients continued treatment until disease progression or unacceptable toxicity. After discontinuation of study drugs, patients were assessed every 3 months up to 1 year for PFS, with visits and/or phone calls.
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Number analyzed (Participants) | 26
months | 4.13 [2.75 to 12.7]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is the percentage of patients whose cancer shrinks or disappears after treatment. Objective response rate was calculated based on the number of patients who had a Complete Response (CR) or a Partial Response (PR). CR and PR were measured according to RECIST v. 1.1 guidelines:
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 9 Cycles (1 cycle = 21 days)
Population: One patient was not evaluable due to non-compliance with capecitabine. Three patients were not evaluable because they did not have 3 cycles of treatment (as required per protocol to be evaluable for efficacy endpoints).
Measure: Number; unit: participants
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Number analyzed (Participants) | 26
participants
  Complete Response | 0
  Partial Response | 4

3. Secondary Outcome: Incidence of Adverse Events
Description: Determine the safety and tolerability of the combination of pembrolizumab and Capecitabine by evaluating the incidence of adverse events. All adverse events will be assessed using the National Cancer Institute Common Terminology Criteria 4.03 criteria (NCI CTCAE 4.03 criteria).
Time Frame: Up to 2 years
Reporting Status: Not Posted

4. Post Hoc Outcome: Clinical Benefit Rate (CBR)
Description: To evaluate the clinical benefit rate (CBR) per RECIST v. 1.1. CBR is the rate of participants with complete response (CR), partial response (PR) or stable disease (SD) > 6 months. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: Up to 14 cycles (1 cycle= 21 days)
Population: One patient was not evaluable due to non-compliance with capecitabine. Patients who received at least one dose of capecitabine and pembrolizumab were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Number analyzed (Participants) | 29
percentage of participants | 28

5. Post Hoc Outcome: 1-year Progression Free Survival (PFS) Rate
Description: To evaluate the 1-year progression free survival (PFS) rate per RECIST v. 1.1.
  PFS is defined as the length of time during and after the treatment that a patient does not experience progression.
  Progressive Disease (PD) as defined per RECIST 1.1 is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  PFS was analyzed using a Kaplan-Meier curve.
Time Frame: Up to 1 year after starting treatment
Population: One patient was excluded from the analysis due to patient non-compliance with capecitabine. Patients who received at least 1 dose of pembrolizumab and capecitabine were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Number analyzed (Participants) | 29
percentage of participants | 20.7

6. Post Hoc Outcome: Median PFS (Median Progression-Free Survival)
Description: as for outcome 1
Time Frame: Approximately 20 months
Population: One patient was not evaluable due to non-compliance with capecitabine. Patients who received at least one dose of pembrolizumab with capecitabine were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Number analyzed (Participants) | 29
months | 4.0 [2.0 to 6.4]

7. Post Hoc Outcome: Objective Response Rate (ORR)
Description: The ORR is the percentage of patients whose cancer shrinks or disappears after treatment. Objective response rate was calculated based on percentage of patients who had a Complete Response (CR) or a Partial Response (PR). CR and PR were measured according to RECIST v. 1.1 guidelines:
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 9 Cycles (1 cycle = 21 days)
Population: One patient was not evaluable due to non-compliance with capecitabine. The analysis included all patients who received at least one dose of capecitabine and pembrolizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment: Pembrolizumab + Capecitabine
Number analyzed (Participants) | 29
percentage of participants | 14

ADVERSE EVENTS:
Time Frame: Patients on study may continue treatment until progression or unacceptable toxicity. AEs currently collected for up to 27 cycles for any patient where one cycle equals 21 days.
Description: Adverse event data shown below includes all events collected and available up until March 30, 2020 for the study. Data collected includes the highest grade of the event experienced for each participant, and thus includes some serious adverse event data.
Arm/Group | Treatment: Pembrolizumab + Capecitabine
All-Cause Mortality (participants affected / at risk) | 17/30
Serious Adverse Events (participants affected / at risk) | 19/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Pembrolizumab + Capecitabine (N=30)
Delerium (Psychiatric disorders) | 1 — Participant also experienced confusion.
Seizure (Nervous system disorders) | 1
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 — One participant also experienced Blood Bilirubin elevated, multi organ failure, CNS progression, AST increased, ALT increased, ALK Phos increased, Hepatitis (Autoimmune), Kidney failure, and Blood bilirubin increased.
Abdominal Pain (Gastrointestinal disorders) | 1
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Other, specify: new bone metastases from primary breast cancer Participant also experienced spinal fracture.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — Participant also experienced chest pain.
Pneumonistis (Respiratory, thoracic and mediastinal disorders) | 1
Blood bilirubin increased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 — Participant also experienced dyspnea.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Pembrolizumab + Capecitabine (N=30)
Anemia (Blood and lymphatic system disorders) | 5
Atrial fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 3
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 4
Hypothyroidism (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 4
Dry eye (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 2
Photophobia (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 15
Dry mouth (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Lip pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 13
Rectal pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 8
Chills (General disorders) | 3
Edema limbs (General disorders) | 6
Fatigue (General disorders) | 13
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Bronchial infection (Infections and infestations) | 1
Lip infection (Infections and infestations) | 2
Papulopustular rash (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 3
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 10
Blood bilirubin increased (Investigations) | 6
Creatinine increased (Investigations) | 1
Fibrinogen decreased (Investigations) | 1
INR increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 7
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 9
Intracranial hemorrhage (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 4
Confusion (Psychiatric disorders) | 4
Delirium (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 5
Acute kidney injury (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 14
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 0
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03044730/Prot_SAP_000.pdf